CLINICAL TRIAL: NCT02052960
Title: Randomized, Controlled, Open Label, Multicenter, Phase II Study to Evaluate the Efficacy and Safety of CetuGEX™ Plus CT in Comparison to Cetuximab Plus CT in Patients With Stage III/IV Recurrent and/or Metastatic SCCHN
Brief Title: CetuGEX™ in Comparison to Cetuximab for the Treatment of Patients With Head and Neck Cancer
Acronym: RESGEX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Glycotope GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEXMab52201; 2013-000931-28 (EudraCT Number)
Record Dates: First submitted 2014-01-27; First posted 2014-02-03 (Estimated); Results first posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Carcinoma, Squamous Cell of Head and Neck
Keywords: tomuzotuximab; cetuximab; SCCHN
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cetuximab; Drug Therapy; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CetuGEX™ plus chemotherapy (Experimental): 720 mg weekly administration
  Interventions: Drug: CetuGEX™; Drug: Chemotherapy
- Cetuximab plus chemotherapy (Active Comparator): 250 mg/m2 weekly administration
  Interventions: Drug: Cetuximab; Drug: Chemotherapy

INTERVENTIONS:
Drug: CetuGEX™ — 60 mg/day 0, 930 mg/day 1, followed by 720 mg i.v. weekly administration
  Other Names: Tomuzotuximab
  Arms: CetuGEX™ plus chemotherapy
Drug: Cetuximab — 400 mg/sqm body surface area (BSA) on day 1, followed by 250 mg/sqm BSA i.v. weekly administration
  Other Names: Erbitux®
  Arms: Cetuximab plus chemotherapy
Drug: Chemotherapy — Combination of Cisplatin and 5-Fluorouracil (Carboplatin may substitute Cisplatin following the 1st cycle of therapy in case of toxicity)
  Other Names: Combination of Cisplatin and 5-Fluorouracil

SUMMARY:
The aim of the study is to evaluate the efficacy of CetuGEX™ for the treatment of patients with stage III/IV recurrent and/or metastatic SCCHN as compared to cetuximab (both in combination with platinum-based chemotherapy) in terms of progression-free survival (PFS).

DETAILED DESCRIPTION:
Indication: First line systemic treatment for stage III/IV recurrent and/or metastatic squamous cell carcinoma of the head and neck (SCCHN)

Primary Objective:

To evaluate the efficacy of CetuGEX™ for the treatment of patients with stage III/IV recurrent and/or metastatic SCCHN as compared to cetuximab (both in combination with platinum-based chemotherapy) in terms of progression-free survival (PFS).

Secondary Objectives:

To evaluate further efficacy criteria, safety and quality of life (QoL) of patients with stage III/IV recurrent and/or metastatic SCCHN treated with CetuGEX™ as compared to cetuximab (both in combination with platinum-based chemotherapy).

To assess pharmacokinetic (PK) parameters and profiles of CetuGEX™. To assess efficacy and safety based on genetic markers for immune response (Fc-gamma receptor [FcγR] allotypes) and biomarkers (exploratory only).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed recurrent and/or metastatic SCCHN not eligible for local treatment.
2. Patients with measurable disease according to RECIST 1.1.
3. Patients aged at least 18 years at screening.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
5. Minimum life expectancy of 3 months.
6. Tissue samples available for specific and therapy-related biological assessments.
7. If female and of childbearing potential, was non-lactating and had negative pregnancy test results at screening and prior to randomization.
8. If female, was either not of childbearing potential (defined as postmenopausal for at least 1 year or surgically sterile [bilateral tubal ligation, bilateral oophorectomy, or hysterectomy]) or willing to use highly effective contraceptives during study participation until 6 months after last administration of any study medication, particularly cisplatin or carboplatin, with a failure rate <1% according to the Note for Guidance on non-clinical safety studies for the conduct of human clinical trials and marketing authorization for pharmaceuticals (CPMP/ICH/286/95) of the European Medicines Agency. Male patients who had partners of childbearing potential had to confirm adequate use of highly effective contraceptives during study participation until 6 months after last administration of any study medication, particularly cisplatin or carboplatin, as well.
9. Willing and able to comply with the protocol.
10. Willing and able to provide written informed consent.

Exclusion Criteria:

1. Prior systemic chemotherapy, except if given as part of a multimodal treatment for locally advanced disease which was completed more than 6 months prior to randomization.
2. Cetuximab or other epidermal growth factor receptor (EGFR)-targeting agent treatment, except if given as part of a multimodal treatment for locally advanced disease which was completed more than 6 months prior to randomization.
3. Surgery (other than minor interventions like diagnostic biopsy or intravenous port implantation) or irradiation within 30 days before randomization.
4. Concomitant antitumor therapy or concomitant immunotherapy, live vaccines including yellow fever vaccination (as per cisplatinum Summary of Product Characteristics [SmPC]).
5. Concomitant corticosteroid treatment unless specified within the protocol.
6. Clinical evidence of brain metastasis or leptomeningeal involvement.
7. Patients with nasopharyngeal tumors.
8. Concomitant malignant disease, except for adequately treated tumors with high likelihood of being cured (e.g., basal cell cancer of the skin, cervical cancer or breast cancer in situ). Patients with previous malignancies but without evidence of disease for at least 5 years were allowed to enter the study.
9. Patients with renal or hepatic impairment (serum creatinine and bilirubin >1.5 fold above the upper limit of normal ranges, creatinine clearance <60 mL/min, and transaminase >5-fold above the upper limit of normal ranges) and patients with hematology parameters outside the normal ranges (hemoglobin <9 g/dL, absolute neutrophil count <1500/mm3 and platelet count <105/mm3) at screening as well as patients with impaired auditory function or platinum-related neuropathy.
10. Clinically active infections ≥Grade 2 using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4 and/or requiring intravenous antibiotics.
11. Known active hepatitis B or C.
12. Known human immunodeficiency virus (HIV) infection.
13. Myocardial infarction within 6 months prior to screening.
14. Symptomatic congestive heart failure (New York Heart Association Grade 3 or 4), unstable angina pectoris within 6 months prior to screening, significant cardiac arrhythmia, history of stroke, or transient ischemic attack within 1 year prior to screening.
15. History of keratitis requiring medical interventions within the last 5 years or interstitial lung disease.
16. Patients with any other disorder that, in the opinion of the investigator, might have interfered with the conduct of the study.
17. Patients with an unstable condition (e.g., psychiatric disorder, a recent history of drug or alcohol abuse, interfering with study compliance, within 6 months prior to screening) or otherwise thought to be unreliable or incapable of complying with the requirements of the protocol.
18. Patients institutionalized by official means or court order.
19. Receipt of any other IMP within the last 30 days before randomization or any previous CetuGEX™ administration.
20. Prior allergic reaction to a monoclonal antibody, grade 3 infusion related reaction (IRR) or any grade 4 reaction to a monoclonal antibody.
21. Known sensitivity to any component of the IMP and medication used in this study.
22. Known dihydropyrimidine dehydrogenase deficiency (France only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2017-08-28 (Actual); Study Completion 2017-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Keilholz, Prof, Principal Investigator — Charite University, Berlin, Germany
Locations (32):
- Belgium (3):
  - Glycotope-contracted Research Facility, Antwerp
  - Glycotope-contracted Research Facility, Brussels
  - Glycotope-contracted Research Facility, Ghent
- France (5):
  - Glycotope-contracted Research Facility, Avignon
  - Glycotope-contracted Research Facility, Lille
  - Glycotope-contracted Research Facility, Lyon
  - Glycotope-contracted Research Facility, Nice
  - Glycotope-contracted Research Facility, Saint-Herblain
- Germany (7):
  - Glycotope-contracted Research Facility, Aachen
  - Glycotope-contracted Research Facility, Berlin
  - Glycotope-contracted Research Facility, Dresden
  - Glycotope-contracted Research Facility, Essen
  - Glycotope-contracted Research Facility, Hamburg
  - Glycotope-contracted Research Facillity, Hanover
  - Glycotope-contracted Research Facility, Leipzig
- Italy (2):
  - Gycotope-contracted Research Facility, Milan
  - Glycotope-contracted Research Facility, Pavia
- Poland (5):
  - Glycotope-contracted Research Facility, Bydgoszcz
  - Glycotope-contracted Research Facility, Krakow
  - Glycotope-contracted Research Facility, Lodz
  - Glycotope-contracted Research Facility, Lublin
  - Glycotope-contracted Research Facility, Warsaw
- Romania (7):
  - Glycotope-contracted Research Facility, Brasov
  - Glycotope-contracted Research Facility, Clui-Napoca
  - Glycotope-contracted Research Facility, Craiova
  - Glycotope-contracted Research Facility, Oradea
  - Glycotope-contracted Research Facility, Ploieşti
  - Glycotope-contracted Research Facility, Timișoara
  - Glycotope-contracteed Research Facility, Timișoara
- Spain (3):
  - Glycotope-contracted Research Facility, Barcelona
  - Glycotope-contracted Research Facility, Madrid
  - Glycotope-contracted Research Facility, Valencia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- CetuGEX in Combination With Chemotherapy: CetuGEX™ was administered as infusion to all patients randomized to the CetuGEX™ arm, once weekly. The initial dose was 990 mg and subsequent doses were 720 mg once weekly. Chemotherapy consisted of 5-FU (1000 mg/m2/d, day 1-4) and cisplatin (100 mg/m2, on day 1).Treatment cycles were scheduled to be repeated every 3 weeks for a maximum of 6 cycles, and followed by a weekly single-agent maintenance therapy of CetuGEX.
- Cetuximab in Combination With Chemotherapy: Cetuximab was administered once weekly as infusion to all patients randomized to the cetuximab arm.The initial dose was 400 mg/m2 body surface area (BSA) and each subsequent dose was 250 mg/m2 BSA. Chemotherapy consisted of 5-FU (1000 mg/m2/d, day 1-4) and cisplatin (100 mg/m2, on day 1).Treatment cycles were scheduled to be repeated every 3 weeks for a maximum of 6 cycles, and followed by a weekly single-agent maintenance therapy of cetuximab.
Period: Overall Study
Arm/Group | CetuGEX in Combination With Chemotherapy | Cetuximab in Combination With Chemotherapy
Started | 117 | 123
Treated Patients (Included all patients who received at least 1 dose of trial medication. This population was used for safety analyses (= Safety Population).) | 115 | 122
Completed | 63 | 77
Not Completed | 54 | 46
Not completed — Adverse Event | 19 | 17
Not completed — Protocol Violation | 4 | 3
Not completed — Withdrawal by Subject | 6 | 11
Not completed — Other | 25 | 15

BASELINE CHARACTERISTICS:
Population: The intention-to-treat (ITT) population consisted of all randomized patients. The ITT population was the primary population for the efficacy analysis. The safety population included all patients who received at least 1 dose of trial medication (N=237). This population was used for safety analyses (adverse events).
Groups:
- Total: Total of all reporting groups
Arm/Group | CetuGEX™ Plus Chemotherapy | Cetuximab Plus Chemotherapy | Total
Number analyzed (Participants) | 117 | 123 | 240
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 88 | 89 | 177
  >=65 years | 29 | 34 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (7.54) | 59.8 (7.91) | 59.8 (7.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 99 | 106 | 205
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Romania | 24 | 19 | 43
  Belgium | 5 | 8 | 13
  Poland | 29 | 29 | 58
  Italy | 1 | 7 | 8
  France | 19 | 25 | 44
  Germany | 33 | 29 | 62
  Spain | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: The primary efficacy endpoint was PFS as assessed by the investigator. Date of disease progression was defined as the date of imaging (based on computed tomography (CT) scans or magnetic resonance imaging (MRI)) showing disease progression, as assessed by the investigator according to adapted immune-related RECIST 1.1 (modified irRC). Disease progression was defined as a 20% increase in tumor burden, taking as reference the smallest tumor burden recorded since the treatment started; confirmation by a second scan was not required. The PFS time was censored at the time of the last tumor assessment if the patient was alive and without progression at the last time of observation.
Time Frame: The PFS was defined as time from randomization until disease progression or death of any cause, up to 24 month
Population: Intent-to-treat-population
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- CetuGEX: CetuGEX™ was administered as infusion to all patients randomized to the CetuGEX™ arm, once weekly. The initial dose was 990 mg and subsequent doses were 720 mg once weekly
- Cetuximab: Cetuximab was administered once weekly as infusion to all patients randomized to the cetuximab arm.The initial dose was 400 mg/m2 body surface area (BSA) and each subsequent dose was 250 mg/m2 BSA.
Arm/Group | CetuGEX | Cetuximab
Number analyzed (Participants) | 117 | 123
weeks | 27.7 [25.3 to 33.7] | 26.4 [24.9 to 31.3]
Statistical Analysis 1: Comparison: CetuGEX vs Cetuximab; Test type: Superiority; p = 0.86, Log Rank; Hazard Ratio (HR) = 1.000, 95% CI 2-sided [0.736 to 1.359]

2. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective response rate is the percentage of patients with a tumor size reduction of a predefined amount for a minimum time period and it is defined as the sum of complete responses (CR) and partial responses (PR).
  CR: Disappearance of all non-nodal target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (< 10 mm short axis).
  PR: At least a 30% decrease in the tumor burden (sum of the longest lesion diameter (LD) of target lesions (including the short axes of any target lymph nodes plus measurable new lesions), taking as reference the baseline sum diameters.
Time Frame: Time from randomization until disease progression or death, whichever occurs first, up to 24 month.
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | CetuGEX | Cetuximab
Number analyzed (Participants) | 117 | 123
Participants | 52 | 57
Statistical Analysis 1: Comparison: CetuGEX vs Cetuximab; Test type: Superiority; p = 0.77, Chi-squared; Mean Difference (Net) = -1.9, 95% CI 2-sided [-14.5 to 10.7]

3. Secondary Outcome: Clinical Benefit Rate
Description: The clinical benefit rate is the percentage of patients with an objective response or stable disease (SD). SD is defined as not meeting criteria of complete response and partial response, in absence of meeting criteria for disease progression. Follow-up measurements must have met the SD criteria at least once after randomization at a minimum interval of 8 weeks.
Time Frame: Time from randomization until disease progression or death, whichever occurs first, up to 24 month.
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | CetuGEX | Cetuximab
Number analyzed (Participants) | 117 | 123
Participants | 88 | 94
Statistical Analysis 1: Comparison: CetuGEX vs Cetuximab; Test type: Superiority; p = 0.83, Chi-squared; Mean Difference (Net) = -1.21, 95% CI 2-sided [-12.05 to 9.63]

4. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure is defined as the time from randomization to treatment discontinuation for any reason, including disease progression, treatment toxicity, patient preference, or death.
Time Frame: Time to treatment failure, defined as the interval between the date of randomization and the date of treatment discontinuation for any reason, up to 24 month.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | CetuGEX | Cetuximab
Number analyzed (Participants) | 116 | 123
weeks | 22.1 [17.0 to 25.7] | 23.3 [16.1 to 25.6]
Statistical Analysis 1: Comparison: CetuGEX vs Cetuximab; Test type: Superiority; p = 0.70, Log Rank; Hazard Ratio (HR) = 1.057, 95% CI 2-sided [0.814 to 1.372]

5. Secondary Outcome: Overall Survival
Description: The overall survival is defined as the duration of time from randomization to the time of death.
Time Frame: Time from randomization to the time of death, up to 24 month.
Population: Intent-to-treat- population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | CetuGEX | Cetuximab
Number analyzed (Participants) | 117 | 123
weeks | 49.7 [40.7 to 73.9] | 59.0 [52.9 to 70.3]
Statistical Analysis 1: Comparison: CetuGEX vs Cetuximab; Test type: Superiority; p = 0.96, Log Rank; Hazard Ratio (HR) = 1.012, 95% CI 2-sided [0.734 to 1.396]

6. Secondary Outcome: Time of Global Health Status Deterioration
Description: Quality of Life (QoL) scores as assessed by European Oncology Research Trials Committee (EORTC) QoL questionnaires (QLQ) EORTC-QLQ-C30.
  Scores are on a scale of 0 to 100, where 100 represents the highest possible QoL.Time to first deterioration of at least 10 points.
Time Frame: From randomization up to end-of study visit, up to 24 month
Population: Intent-to treat population. 158 patients were evaluable for this Outcome Measure.
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | CetuGEX in Combination With Chemotherapy | Cetuximab in Combination With Chemotherapy
Number analyzed (Participants) | 76 | 82
weeks | 43.4 [14.0 to 61.4] | 31.3 [11.7 to 63.0]

ADVERSE EVENTS:
Time Frame: up to 24 month
Arm/Group | CetuGEX | Cetuximab
All-Cause Mortality (participants affected / at risk) | 20/115 | 14/122
Serious Adverse Events (participants affected / at risk) | 70/115 | 78/122
Other Adverse Events (participants affected / at risk) | 114/115 | 121/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CetuGEX (N=115) | Cetuximab (N=122)
Hypotension (Vascular disorders) | 3 | 2
Blood creatinine increased (Investigations) | 2 | 3
Myocardial infarction (Cardiac disorders) | 2 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Anemia (Blood and lymphatic system disorders) | 9 | 9
Neutropenia (Blood and lymphatic system disorders) | 8 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 2
Leucopenia (Blood and lymphatic system disorders) | 1 | 4
Cerebrovascular accident (Nervous system disorders) | 2 | 1
General physical health deterioration (General disorders) | 2 | 2
Device dislocation (General disorders) | 1 | 2
Fatigue (General disorders) | 2 | 1
Mucosal inflammation (General disorders) | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 2
Nausea (Gastrointestinal disorders) | 3 | 2
Vomiting (Gastrointestinal disorders) | 2 | 2
Renal failure (Renal and urinary disorders) | 2 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 4 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 4
Decreased appetite (Metabolism and nutrition disorders) | 2 | 3
Pneumonia (Infections and infestations) | 12 | 9
Sepsis (Infections and infestations) | 3 | 7
Device related infection (Infections and infestations) | 5 | 4
Lung abscess (Infections and infestations) | 0 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CetuGEX (N=115) | Cetuximab (N=122)
Hypotension (Vascular disorders) | 16 (20) | 16 (24)
Hypertension (Vascular disorders) | 11 (30) | 8 (13)
Fatigue (General disorders) | 41 (82) | 38 (81)
Asthenia (General disorders) | 34 (60) | 37 (75)
Mucosal inflammation (General disorders) | 24 (45) | 36 (63)
Pyrexia (General disorders) | 16 (17) | 24 (30)
Chills (General disorders) | 26 (28) | 6 (6)
General physical health deterioration (General disorders) | 7 (10) | 6 (6)
Pulmonary embolism (Psychiatric disorders) | 8 (13) | 4 (5)
Weight decreased (Investigations) | 42 (83) | 39 (72)
Blood creatinine increased (Investigations) | 11 (19) | 8 (15)
Platelet count decreased (Investigations) | 7 (13) | 6 (6)
Tachycardia (Cardiac disorders) | 10 (11) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 44 (104) | 56 (152)
Neutropenia (Blood and lymphatic system disorders) | 47 (105) | 51 (124)
Leukopenia (Blood and lymphatic system disorders) | 33 (98) | 37 (90)
Thrombocytopenia (Blood and lymphatic system disorders) | 21 (48) | 26 (69)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 15 (21)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (17) | 14 (16)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 10 (13)
Dizziness (Nervous system disorders) | 14 (16) | 15 (20)
Headache (Nervous system disorders) | 13 (16) | 13 (19)
Neuropathy periphera (Nervous system disorders) | 3 (4) | 9 (19)
Conjunctivitis (Eye disorders) | 10 (16) | 9 (12)
Vertigo (Ear and labyrinth disorders) | 11 (13) | 12 (12)
Tinnitus (Ear and labyrinth disorders) | 8 (10) | 6 (7)
Hearing impaired (Ear and labyrinth disorders) | 6 (6) | 7 (8)
Nausea (Gastrointestinal disorders) | 58 (122) | 63 (162)
Diarrhoea (Gastrointestinal disorders) | 38 (73) | 41 (84)
Vomiting (Gastrointestinal disorders) | 35 (67) | 41 (83)
Constipation (Gastrointestinal disorders) | 34 (47) | 23 (40)
Stomatitis (Gastrointestinal disorders) | 26 (66) | 12 (21)
Dysphagia (Gastrointestinal disorders) | 15 (20) | 16 (22)
Dyspepsia (Gastrointestinal disorders) | 15 (23) | 13 (19)
Abdominal pain (Gastrointestinal disorders) | 7 (17) | 12 (13)
Abdominal pain upper (Gastrointestinal disorders) | 9 (11) | 6 (6)
Renal failure (Renal and urinary disorders) | 5 (7) | 11 (16)
Rash (Skin and subcutaneous tissue disorders) | 44 (116) | 47 (127)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 30 (106) | 21 (64)
Dry skin (Skin and subcutaneous tissue disorders) | 20 (23) | 23 (26)
Skin fissures (Skin and subcutaneous tissue disorders) | 19 (38) | 17 (36)
Acne (Skin and subcutaneous tissue disorders) | 10 (23) | 11 (40)
Alopecia (Skin and subcutaneous tissue disorders) | 9 (10) | 11 (13)
Erythema (Skin and subcutaneous tissue disorders) | 8 (8) | 8 (10)
Pruritus (Skin and subcutaneous tissue disorders) | 10 (16) | 4 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (9) | 7 (8)
Hypomagnesaemia (Metabolism and nutrition disorders) | 53 (146) | 51 (181)
Decreased appetite (Metabolism and nutrition disorders) | 36 (47) | 30 (48)
Hypokalaemia (Metabolism and nutrition disorders) | 20 (35) | 22 (53)
Dehydration (Metabolism and nutrition disorders) | 10 (11) | 13 (14)
Hypocalcaemia (Metabolism and nutrition disorders) | 10 (19) | 13 (20)
Hyponatraemia (Metabolism and nutrition disorders) | 11 (14) | 9 (9)
Paronychia (Infections and infestations) | 16 (36) | 12 (19)
Pneumonia (Infections and infestations) | 13 (17) | 12 (14)
Urinary tract infection (Infections and infestations) | 7 (12) | 6 (7)
Bronchitis (Infections and infestations) | 3 (3) | 9 (14)
Device related infection (Infections and infestations) | 8 (8) | 4 (5)
Sepsis (Infections and infestations) | 4 (4) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication, presentation or use of the methods and/or results of the clinical trial are not permitted without prior written sponsor´s consent.

DOCUMENTS (2):
  • Study Protocol (2015-02-06): https://cdn.clinicaltrials.gov/large-docs/60/NCT02052960/Prot_000.pdf
  • Statistical Analysis Plan (2016-12-21): https://cdn.clinicaltrials.gov/large-docs/60/NCT02052960/SAP_001.pdf